CLINICAL TRIAL: NCT03883672
Title: Study of the Role of Socio-psychological Factors in the Hematopoietic Stem Cell Transplantation Process in People With Hemopathies
Brief Title: Socio-psychological Factors Involved in the Hematopoietic Stem Cell Transplantation Process in People With Hemopathies
Acronym: Psy-Greffe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Principal Investigator, Régis Peffault de Latour, Professor Regis Peffault De Latour, Saint-Louis Hospital, Paris, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AGRAH1
Record Dates: First submitted 2018-12-05; First posted 2019-03-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hematopoietic stem cell transplantation (Experimental): Personality and transactional factors involved in the process and outcomes of hematopoietic stem cell transplantation
  Interventions: Behavioral: Personality and transactional factors

INTERVENTIONS:
Behavioral: Personality and transactional factors — 1. Pre-admission transplant questionnaire: given and collected by the transplant physician during the pre-graft consultation before entering hospitalization (approximatively 15 days before). To be completed by the patient on site (approximately 45 minutes to complete the questionnaire)
  2. Transplant admission questionnaire: given during the first days of hospitalization. To be completed within 6 days and returned to the transplant physician (approximately 30 minutes to complete the questionnaire)
  3. Post-transplant follow-up questionnaire: given in consultation at 6 months by the transplant physician (between 30 and 45 minutes to complete the questionnaire in consultation)

SUMMARY:
Identify the psychological factors (i.e. personality and transactional factors), beneficial and deleterious, at different phases of the transplant process, on the patient's mental health (quality of life, short and long-term post-transplant recovery) and physical health (e.g. infections, relapse, length of hospitalization or even death).

DETAILED DESCRIPTION:
To reach the research purposes, questionnaires will be given to patients at different times during the transplant process :

1. Pre-admission transplant questionnaire: given and collected by the transplant physician during the pre-graft consultation before entering hospitalization (approximatively 15 days before). To be completed by the patient on site (approximately 45 minutes to complete the questionnaire)
2. Transplant admission questionnaire: given during the first days of hospitalization. To be completed within 6 days and returned to the transplant physician (approximately 30 minutes to complete the questionnaire)
3. Post-transplant follow-up questionnaire: given in consultation at 6 months by the transplant physician (between 30 and 45 minutes to complete the questionnaire in consultation)

The questionnaires include validated and standardized scales.

The first questionnaire contains scales on dispositional factors (i.e. personality factors) . The second one is on the so-called transactional adjustment factors. And the third is on post-transplant factors (e. g. post-traumatic growth). Scales from the first and second questionnaire will be used to obtain a longitudinal view.

The study population concerns all patients going to receive an allograft transplantation, aged over 18 years, who have consented to answer the various questionnaires over a period of approximately 7 months . The participants come from the hematology departments of the Saint-Louis Hospital in Paris, the Estaing University Hospital in Clermont-Ferrand and the Brabois Hospital in Nancy.

ELIGIBILITY:
Inclusion Criteria:

* patient with hematopathy with allograft HSC indication
* allograft protocol
* patient over 18 years of age
* patient who has read and understood the information note and who has consented has not objected to participating in the research
* patient affiliated to a social security system (beneficiary )

Exclusion Criteria:

* patients receiving autograft
* patient under 18 years of age
* patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Five Facets Mindfulness Questionnaire (FFMQ) | 15 days before hospitalization
  Assessement of Mindfulness level as a dispositional dimension. Baert et al., 2006 ; Heeren et al., 2011 39-items scale 5 underscores for each facets of mindful trait: to observe (8 items, max=40), to describe (8 items, max= 40), to act with awareness (8 items, max= 40), to non judge (8 items, max= 40, to non react (7 items, max= 35) Range for full scale: [39-195] More the score is high more the mindfulness level is high. No pathological score
General Self Efficacy Scale (GSES) | 15 days before hospitalization
  Assessment of Perceived Self Efficacy level (e.g. Am I think myself able to do something ?) Schwarzer & Jerusalem, 1995 10-items scale. The total score is the sum of all items. Range for full scale : [10-40] More the score is high more the general self efficacy level is high. No pathological score
Authentic sustainable happiness scale (ASHS) | 15 days before hospitalization
  Dambrun et al. (2012) Assessment of a happiness component through 13 items (e.g.: satisfaction, general well-being, serenity, etc.). 2 happiness subscales to sum for obtain the total score of hapiness: "contentment" (8 items) and "inner peace" (5 items). Range for full scale: [13-91]. Range for "contentment subscale": [8-56]. range for "inner peace" subscale: [5-35]. More the score is high, more the level of authentic and sustainable happiness is high. No pathological score.
  Dambrun et al., 2012 16-items scale
Authentic sustainable happiness scale (ASHS) | 6 months after hospitalization
  Dambrun et al. (2012) Assessment of a happiness component through 13 items (e.g.: satisfaction, general well-being, serenity, etc.). 2 happiness subscales to sum for obtain the total score of hapiness: "contentment" (8 items) and "inner peace" (5 items). Range for full scale: [13-91]. Range for "contentment subscale": [8-56]. range for "inner peace" subscale: [5-35]. More the score is high, more the level of authentic and sustainable happiness is high. No pathological score.
  Dambrun et al., 2012 16-items scale
Life Orientation Test-Revised (LOT-R) | 15 days before hospitalization
  Assessment of dispositional Optimism level Scheier, Carver & Bridge,1994 10-items scale: 6 items assessing optimism component and 4 fillers. The total score is the sum of the 6 items. Range for the total scale: [6-42]. More the score is high, more the optimism level is high. No pathological score.
Adult Dispositional Hope Scale (ADHS) | 15 days before hospitalization
  Assessement of Dispositional Hope level of people. Snyder et al., 1991 ; Gana et al., 2012 12-items scale. range for the full scale: [8-64]. 2 subscales: "agency" (4 items, [4-32]), "pathways" (4 items, [4-32]) and 4 fillers. The total score is the sum of the 8 items. More the score is high, more the dispositional hope level is high. No pathological score.
Acceptance and Action Questionnaire-version 2 (AAQ-II) | 15 days before hospitalization
  Assessement of two dimensions of psychological flexibility (involved in a good mental health) Bond et al., 2011 ; Monestès et al., 2009 10-items scale. Range for the full scale [10-70]. The total score is the sum of the 10 items. More the the score is high, more the psychological flexibility is high. No pathological score
Single Item Self Esteem (SISE) | 15 days before hospitalization
  Assessment of self-esteem dimension Robins et al., 2001
  1-item scale. Range of the item [1-7]. More the score is high, more the self-esteem level is high. No pathological score.
Ego Resiliency Scale-revised (EGO-R-r) | 15 days before hospitalization
  Assessment of Resiliency as a dispositional dimension. 2 subscales: "optimal regulation" (6 items, [6-42] and "openness to life experience" (4 items, [4-28]). Range for the full scale: [10-70]. The total score is the sum of the 2 subscales scores (10 items). More the score is high, more the resiliency level is high. No pathological score.
  Alessandri, Vecchione, Caprara, & Letzring, 2011 10-items scale
Avoidance and Fusion Questionnaire for Adults (AFQ) | 15 days before hospitalization
  Assessement of experiential avoidance and fusion, 2 dimensions of psychological inflexibility (involved in the maintenance of emotional disorders as depression or anxiety) Fergus et al., 2012 17-items scale. Range for the full scale: [0-68]. The total score is the sum of the 17 items. More the score is high, more the psychological inflexibility is high. No pathological score
Hospital Anxiety and Depression Scale | 15 days before hospitalization
  Assessement of anxiety and depression symptoms for hospitalized people Zigmond & Snaith, 1983 14-items scale 2 underscores: "depression" score (7 items) and "anxiety" score (7 items). One score for depression is computed (sum of 7 items, [0-21] and one for "anxiety" is computed too (sum of 7 items, [0-21]). For each subscales: a score under 7 is not pathological; between 8 and 10 there is a suspicion of symptomatology; and beyond 11 means an established symptomatology.
Hospital Anxiety and Depression Scale | 6 months after hospitalization
  Assessement of anxiety and depression symptoms for hospitalized people Zigmond & Snaith, 1983 14-items scale 2 underscores: "depression" score (7 items) and "anxiety" score (7 items). One score for depression is computed (sum of 7 items, [0-21] and one for "anxiety" is computed too (sum of 7 items, [0-21]). For each subscales: a score under 7 is not pathological; between 8 and 10 there is a suspicion of symptomatology; and beyond 11 means an established symptomatology.
Toronto Alexithymia Scale-20 (TAS-20) | 15 days before hospitalization
  Assessment of alexithymia level (i.e. difficulties in experiencing and expressing feelings) Bagby, Parker & Taylor, 2003 ; Loas et al., 1997 20-items scale. Range for the full scale: [20-100]. 3 subscales: "difficulty identifying feelings" (7 items, [7-35]), "difficulty describing feelings to others" (5 items, [5-25]), "externally oriented thinking" (8 items, [8-40]). A score beyond 61 is considered as pathological.
Positive Affect and Negative Affect Schedule (PANAS) | 15 days before hospitalization
  Assessment of positive affectivity (curious, motivated, enthusiastic, proud, etc.) and negative affectivity (guilty, nervous, anguished,etc.) levels Watson, Clark & Tellegen, 1988 ; Caci & Baylé, 2007 20-items scale. 2 underscores: positive affectivity score (10 items, [10-50]) and negative affectivity score (10 items, [10-50]). More the score is high for each subscale, more the experience of positive/ negative affectivity is high. No pathological score.
Big Five Inventory (BFI) | 15 days before hospitalization
  Assessment of 5 personality dimensions: extraversion (8 items, [8-40], openness (10 items, [10-50]), consciousness (9 items, [9-45]), agreeableness (8 items, [8-40]) and neuroticism (8 items, [8-40]).
  John & Srivastava, 1999 ; Plaisant et al., 2010 45-items scale 5 underscores for each personality facet. More the score is high for each personality facet, more the level of extraversion/ openness/ consciousness/ agreeableness/neuroticism is high. No pathological score.
Body boundaries scale (BBS) | 15 days before hospitalization
  Assessment of perceived boundaries of body: prominent boundaries or not prominent boundaries are the two extremes of the continuum Dambrun & Ricard, 2012 Analogic scale. range for the full scale [0-15]. More the score is high more the body boundaries are prominent. No pathological score.
General Questionnaire SF-12: mental and social quality of life | 15 days before hospitalization
  Mental and social quality of life assessment 12-items scale. For each item one standardized score of mental and social quality of life is computed ( [5,89058 ; 71,96825])and one standardized score is computed for the physical quality of life ([9,94738 ; 70,02246]). the mean among the general population is 50. More the score is high, more the level of quality of life is high.
General Questionnaire SF-12: mental and social quality of life | 6 months after hospitalization
  Mental and social quality of life assessment 12-items scale. For each item one standardized score of mental and social quality of life is computed ( [5,89058 ; 71,96825])and one standardized score is computed for the physical quality of life ([9,94738 ; 70,02246]). the mean among the general population is 50. More the score is high, more the level of quality of life is high
Social Provisions scale revised | At the 7th day of hospitalization
  Perceived social support assessment in different settings (attachment, reliable alliance, social integration, reassurance of worth, guidance, ...) Cutrona & Russel, 1987 24-items scale. Range for the full scale [16-96]. 4 items for each subscale (range for each subscales: [4-16]). The total score is the sum of all subscales scores. More the score is high, more the social support is high. No pathological score.
Perceived Stress Scale (PSS) | At the 7th day of hospitalization
  Assessement of perceived stress level (i.e. How much life situations are threatening, unpredictable and uncontrollable).
  Cohen, Karmack, Mermelstein, 1983 10-items scale. range for the full scale: [0-40]. The total score is the sum of all the 10 items. Between 0 and 13: low level of perceived stress. Between 14 and 26: middle level of perceived stress. Between 27and 40: high level of perceived stress.
Mental Adjustment to Cancer Scale (MACs) | At the 7th day of hospitalization
  Coping strategies assessment (i.e. What kind of behavioral or emotional strategies are put in place to cope with stressful events). 5 strategies assessed: fighting spirit, avoidance, helplessness-hopelessness, anxious preoccupations, denial.
  Watson et al., 1998 ; Cayrou et al., 2003 45-items scale. For each strategy a score is computed: fighting spirit ([13;52], 14 items), avoidance ([5; 20], 5 items), helplessness-hopelessness ([11;44] ,11 items), anxious preoccupations ([12; 48],12 items), denial ([3; 12], 3 items). More the score is high for each subscale, more the fighting spirit / avoidance/ helplessness-hopelessness/ anxious preoccupations/ denial strategy is used. No pathological score
Mental Adjustment to Cancer Scale (MACs) | 6 months after hospitalization
  Coping strategies assessment (i.e. What kind of behavioral or emotional strategies are put in place to cope with stressful events). 5 strategies assessed: fighting spirit, avoidance, helplessness-hopelessness, anxious preoccupations, denial.
  Watson et al., 1998 ; Cayrou et al., 2003 45-items scale. For each strategy a score is computed: fighting spirit ([13;52], 14 items), avoidance ([5; 20], 5 items), helplessness-hopelessness ([11;44] ,11 items), anxious preoccupations ([12; 48],12 items), denial ([3; 12], 3 items). More the score is high for each subscale, more the fighting spirit / avoidance/ helplessness-hopelessness/ anxious preoccupations/ denial strategy is used. No pathological score
Levenson scale - Internality- Power of others and Hasard scale (IPAH scale ) | At the 7th day of hospitalization
  Assessment of 3 locus of control facets : Internality; externality (power of others); externality (chance). This scale aims to determine to whom or what do individuals attribute the reasons for the occurrence of an event.
  Jutras, 1987 24-items scale. 3 underscores are computed: internality score (8 items, [6-48]), externality/ power of others (8 items, [6-48]) and externality/ hasard (8 items, [6-48]). More the score for each subscale is high more the internality / externality level is high. No pathological score.
Brief Strengths Test | At the 7th day of hospitalization
  Assessement of personal strengths involved in resiliency, good mental health, happiness. Clustered in 6 different virtues : wisdom and knowledge, courage, humanity, justice, temperance, transcendence.
  Park, Peterson & Seligman, 2004 24-items scale. range for the full scale: [24-120]. 6 underscores are computed for each virtue: wisdom and knowledge (5 items, [5-25]), courage (4 items, [4-20]), humanity (3 items, [3-15]), justice (3 items, [3-15]), temperance (4 items, [4-20]), transcendence (5 items, [5-25]). More the score is high, more the level of wisdom and knowledge/ courage/ humanity/ justice/ temperance/ transcendence is high. No pathological score.
Brief Strengths Test | 6 months after hospitalization
  Assessement of personal strengths involved in resiliency, good mental health, happiness. Clustered in 6 different virtues : wisdom and knowledge, courage, humanity, justice, temperance, transcendence.
  Park, Peterson & Seligman, 2004 24-items scale. range for the full scale: [24-120]. 6 underscores are computed for each virtue: wisdom and knowledge (5 items, [5-25]), courage (4 items, [4-20]), humanity (3 items, [3-15]), justice (3 items, [3-15]), temperance (4 items, [4-20]), transcendence (5 items, [5-25]). More the score is high, more the level of wisdom and knowledge/ courage/ humanity/ justice/ temperance/ transcendence is high. No pathological score.
Positive orientation to others scale | At the 7th day of hospitalization
  Assessment of positive orientation to others level. Braithwaite & Law, 1985 13-items scale. range for the full scale: [13-91]. The total score is the sum of the 13 items. More the score is high, more the orientation to others level is high. No pathological score
Positive orientation to others scale | 6 months after hospitalization
  Assessment of positive orientation to others level. Braithwaite & Law, 1985 13-items scale. range for the full scale: [13-91]. The total score is the sum of the 13 items. More the score is high, more the orientation to others level is high. No pathological score
Intrinsic spirituality scale | At the 7th day of hospitalization
  Assessment of spirituality dimension. How much people think spirituality is important for them? Hodge, 2003 6-items scale. Range for the full scale: [0-60]. The total score is the sum of the 6 items. More the score is high, more the intrinsic spirituality level is high. No pathological score
Intrinsic spirituality scale | 6 months after hospitalization
  Assessment of spirituality dimension. How much people think spirituality is important for them? Hodge, 2003 6-items scale. Range for the full scale: [0-60]. The total score is the sum of the 6 items. More the score is high, more the intrinsic spirituality level is high. No pathological score
Satisfaction with Life Scale | At the 7th day of hospitalization
  Assessment of cognitive component of happiness. This is a general assessment of people life.
  Diener et al.,1985 5-items scale. Range for the full scale: [5-35]. [5-9] : extremely dissatisfied; [10-14]: dissatisfied; [15-19]: slightly dissatisfied; 20: neutral; [21-25]: slightly satisfied; [26-30]: satisfied; [31-35]: extremely satisfied.
Satisfaction with Life Scale | 6 months after hospitalization
  Assessment of cognitive component of happiness. This is a general assessment of people life.
  Diener et al.,1985 5-items scale. Range for the full scale: [5-35]. [5-9] : extremely dissatisfied; [10-14]: dissatisfied; [15-19]: slightly dissatisfied; 20: neutral; [21-25]: slightly satisfied; [26-30]: satisfied; [31-35]: extremely satisfied.
Personal Growth scale | At the 7th day of hospitalization
  Assessment of one dimension of psychological well-being. Ryff & Essex, 1992 14-items scale. range for the full scale: [14-84]. Total score is the sum of the 14 items. More the score is high, more the level of personal growth is high. No pathological score.
Personal Growth scale | 6 months after hospitalization
  Assessment of one dimension of psychological well-being. Ryff & Essex, 1992 14-items scale. range for the full scale: [14-84]. Total score is the sum of the 14 items. More the score is high, more the level of personal growth is high. No pathological score.
Post Traumatic Growth Inventory | 6 months after hospitalization
  Assessment of post traumatic growth level which encountered with traumatized people. 5 different dimensions of PTG: changes in relationships , spirituality , personal growth , personal strength, new possibilities, life satisfaction.
  Tedeschi & Calhoun, 2004 ; Cadell, Suarez & Hemsworth, 2015 21-items scale. range for the full scale: [0-105]. The total is the sum of the 21 items 5 underscores are computed: changes in relationships (7 items, [0-35]) , spirituality (2 items, [0-10]) , personal strength (4 items, [0-20]), new possibilities (5 items, [0-25]),life satisfaction (3 items, [0-15]). More the score is high, more the level of post traumatic growth is high. No pathological score.
Stress version of post traumatic stress disorder scale | 6 months after hospitalization
  Assessment of traumatism level and traumatic symptomatology (e.g. repetition of traumatic event)Weathers et al., 1993 17-items scale. Range for the full scale: [17-85]. The total is the sum of the 17 items. 3 underscores are computed: "repetition of the traumatic event" (5 items, [5-25]), "avoidance" (7 items, [5-35]), "neurovegetative hyperactivity" (5 items, [5-25]). A score beyond 44 is considered as pathological score.
Socio-demographic informations: Age | 15 days before hospitalization
  year
Socio-demographic informations: sex | 15 days before hospitalization
  2 propositions: man or woman
Socio-demographic informations: marital status | 15 days before hospitalization
  5 propositions; single, couple, married, widowed, other
Socio-demographic informations: country | 15 days before hospitalization
  people note the country where they were born
Socio-demographic informations: educational level | 15 days before hospitalization
  What level of education (i.e. degree)
Socio-demographic informations: socioprofessional category | 15 days before hospitalization
  what a job it is
Socio-demographic informations: religion | 15 days before hospitalization
  2 propositions: YES or NO
complementary informations: weight | 15 days before hospitalization
  they indicate it in kilograms
complementary informations: size | 15 days before hospitalization
  they indicate it in meter and centimeters
complementary informations: sleeping hours | 15 days before hospitalization
  they indicate it in number of sleeping hours for each night
complementary informations: alcohol consumption | 15 days before hospitalization
  2 propositions: YES or NO
complementary informations: cigarette consumption | 15 days before hospitalization
  2 propositions: YES or NO
complementary informations: physical activity | 15 days before hospitalization
  2 propositions: YES or NO
complementary informations: artistic activity | 15 days before hospitalization
  2 propositions: YES or NO
complementary informations: dietary regime | 15 days before hospitalization
  2 propositions: YES or NO
Physical health informations (PROMISE database) | 7 months after hospitalization
  All these informations are extracted from PROMISE database : type and stage of hemopathy, type of conditioning (myeloablative, non-myeloablative). During follow-up, transplant intake, acute and chronic GvHD, infections, number of days in hospital, relapse and death (and cause)

CONTACTS AND LOCATIONS:
Overall Officials: Régis Peffault De Latour, Pr., Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (1):
- Régis Peffault De Latour, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corman M, Rubio MT, Cabrespine A, Brindel I, Bay JO, De La Tour RP, Dambrun M. Retrospective and prospective measures of post-traumatic growth reflect different processes: longitudinal evidence of greater decline than growth following a hematopoietic stem-cell transplantation. BMC Psychiatry. 2021 Jan 11;21(1):27. doi: 10.1186/s12888-020-03007-y. PMID 33430807